CLINICAL TRIAL: NCT04344652
Title: Prospective Evaluation of a Smartphone Application, GoCheckKids TM, as a Screening Tool for Leukocoria in the Infant and Pediatric Population
Brief Title: Photoscreening for Retinoblastoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study administratively closed at IRB prior to enrollment.
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AR01
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2020-04

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Intervention Model Description: Single visit cross sectional prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Photoscreening (Experimental): Photoscreening of patients 0 to 10 years of age
  Interventions: Device: Photoscreening -

INTERVENTIONS:
Device: Photoscreening - — external picture taken with a an phone based app

SUMMARY:
Retinoblastoma is the most common pediatric eye malignancy and manifests between 1 and 5 years of age. The tumor is most often diagnosed by leukocoria ( white reflex in the pupil). There is often a significant delay in diagnosis and early diagnosis enables good life prognosis and better vision outcome.There is currently not a standardized screening protocol for detection of retinoblastoma. Vision screening methods are recommended for children 3-5 years of age. The investigators are attempting to use instrument based screening started from birth to detect leukocoria.

ELIGIBILITY:
Inclusion Criteria:

* Age birth to 10 years
* Informed consent given by parent or legal guardian

Exclusion Criteria:

* None

Ages: 0 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Reliability to detect leukocoria | 1 year
  Testing the reliability of the app to detect leukocoria with good sensitivity and specificity

IPD SHARING:
Plan to Share IPD: No